CLINICAL TRIAL: NCT04953260
Title: Comparative Study of Advance Platelet Rich Fibrin/Concentrated Growth Factor Technology in Regenerative Periodontal Surgery: a Randomized Controlled Clinical Trial
Brief Title: Comparative Study of APRF/CGF Technology in GTR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2020-1021
Record Dates: First submitted 2021-01-11; First posted 2021-07-07 (Actual); Last update posted 2021-07-07 (Actual); Status verified 2021-01

CONDITIONS: Chronic Periodontitis; Intrabony Periodontal Defect
Keywords: guided tissue regeneration; APRF; CGF; Intrabony defect; Chronic periodontitis
MeSH Terms: conditions — Chronic Periodontitis

STUDY DESIGN:
Intervention Model Description: This study is a single-center, simple, randomized parallel group design clinical trial in which each random group is allocated according to the proportion of 1:1:1
Who Masked: Investigator, Outcomes Assessor
Masking Description: Researcher B is responsible for including the subjects and assigning the number of the subjects according to the order of treatment. During the operation, researcher B will give the sealed envelope to the surgeon L according to the number, then leave, and will not participate in surgery, measurement and other studies. Researcher C is responsible for measuring various indicators on a regular basis. Until the end of the experiment, C did not know the grouping of the subjects.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- GTR group (No Intervention): only conventional GTR technique was used to treat periodontal bone defect,
- APRF+GTR group (Active Comparator): GTR technique combined with APRF was used to treat periodontal bone defect
  Interventions: Other: APRF
- CGF+GTR group (Active Comparator): GTR technique combined with CGF was used to treat periodontal bone defect
  Interventions: Other: CGF

INTERVENTIONS:
Other: APRF — 20ml venous blood was collected from the elbow before operation and centrifuged with a special centrifuge. One piece of APRF gel was chopped and mixed with Bio-oss, and the other piece was pressed into a thin film; the mixture of APRF and Bio-oss was filled into the bone defect, covered with a properly trimmed Bio-gide film, and then covered with APRF film
  Arms: APRF+GTR group
Other: CGF — 20ml venous blood was collected from the elbow before operation and centrifuged with a special centrifuge. One piece of CGF gel was chopped and mixed with Bio-oss, and the other piece was pressed into a thin film; the mixture of CGF and Bio-oss was filled into the bone defect, covered with a properly trimmed Bio-gide film, and then covered with CGF film
  Arms: CGF+GTR group

SUMMARY:
Guided tissue regeneration(GTR) uses membranous materials to shield gingival epithelial cells and connective tissue cells which grow more rapidly, creating an effective closed space and time for periodontal ligament cells with regenerative potential, so that new cementum is formed on the root surface and periodontal ligament fibers are embedded, resulting in regenerative healing. In order to improve the effect of periodontal regeneration therapy, as early as 1990s, scholars began to mix platelet concentrate and bone graft in periodontal regenerative surgery to improve the ability of local bone induction and tissue healing. Studies have shown that platelet concentrate, which is rich in a variety of growth factors in autologous blood, can promote soft tissue and bone tissue healing by acting on tissue healing cells (osteoblasts, epithelial cells, connective tissue cells, etc.). It is closely related to periodontal regeneration; the regenerative component of platelet concentrate, growth factor, and the structure of fibrin network containing growth factor are the key to promote tissue repair and regeneration.Modified platelet-rich fibrin (advanced platelet rich fibrin,APRF) and concentrated growth factor (CGF) are the latest generation of platelet concentrates. A number of studies have shown that APRF and CGF contain more cytokines, have a denser fibrin network, and show stronger ability to promote the migration and proliferation of gingival fibroblasts, suggesting that both of them may have better ability to promote bone tissue healing. At present, the latest generation of platelet concentrate has been widely used in implant surgery, but their clinical effects in periodontal regeneration surgery are still lack of conclusive evidence. there is no report on comparing the clinical effects of the two through randomized clinical controlled trials.

ELIGIBILITY:
Inclusion Criteria:

1. The age of the patient is 18-80 years old.
2. selection of affected teeth: there is still at least one site of periodontal probing depth ((PD) ≥ 5mm) at 6-8 weeks after initial periodontal treatment,and the degree of mobility is less than grade II or II-III degree but without mobility after fixation.Imaging evaluation shows that the tooth has a Intrabony defect which is larger than 3mm, and there is no history of periodontal surgery at this site, and the affected tooth has no obvious symptoms of discomfort.
3. The patient has good compliance, good plaque control after basic treatment (bleeding index and plaque index < 20%). He/She can understand the purpose of the test and is willing to cooperate with surgical treatment and follow-up. He/She voluntarily participates in the trial and signs informed consent.

Exclusion Criteria:

1. In the past 6 months, patients who chewed smokeless tobacco, smoked a pipe or cigar once a week, or smoked more than 20 cigarettes per week (1 pack per week);
2. Patients took any drug affecting platelet function or had a platelet count less than 200000/mm3 3 months before blood collection.
3. Patients have taken antiepileptic drugs, antihistamines, antidepressants, sedatives, sedatives, anti-inflammatory drugs or daily analgesics within 1 month before operation;
4. Patients with a history of diabetes or patients with abnormal blood glucose test (fasting blood glucose ≥ 7mmol/L);
5. Liver and renal dysfunction (AST, ALT ≥ 1.5 times ULN, creatinine ≥ 1.5 times ULN);
6. Patients with severe endocrine and metabolic diseases.
7. Those with a history of grade 3 hypertension;
8. Those with a history of osteoporosis;
9. Those with a history of autoimmune diseases;
10. Those with a history of malignant tumor or other serious diseases who are not suitable for surgery or cause observation of tooth loss;
11. Pregnant or lactating women;
12. Patients with local anesthetic allergy.
13. Clinical or radiological findings showed acute infection, apical lesions, root fractures, severe root deformities, cementum beads, indelible enamel protuberances, untreated caries at the enamel or root boundary, and restoration reaching subgingival and/or below CEJ or marginal incongruity
14. All kinds of subjects who can cause artifacts in oral imaging examination, such as: the study teeth and their adjacent teeth are metal dentures and porcelain teeth;
15. The affected teeth have root furcation lesions

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2020-08-25 (Actual); Primary Completion 2022-03 (Estimated); Study Completion 2022-03 (Estimated)

PRIMARY OUTCOMES:
CAL (clinical attachment level) | Baseline(V0)，Change from Baseline at 12 weeks (V1)，Change from Baseline at 24 weeks (V2)，Change from Baseline at 48 weeks (V3)
  The distance from periodontal pocket bottom to CEJ was measured by periodontal probe (mm). Record six sites of each tooth (the mesial, median and distal site of the buccal and tongue surface ).In order to ensure the operability and scientificity of follow-up, it is defined as follows.

SECONDARY OUTCOMES:
PD（probe depth） | Baseline(V0)，Change from Baseline at 12 weeks (V1)，Change from Baseline at 24 weeks (V2)，Change from Baseline at 48 weeks (V3)
  use a periodontal probe (UNC-15,Hu-Friedy,Chicago,IL) paralleling to the long axis of the tooth to measure the distance from the bottom of the periodontal pocket to the gingival margin (mm), record six sites of each tooth (the mesial, median and distal site of the buccal and tongue surface ).
mobility | Baseline(V0)，Change from Baseline at 12 weeks (V1)，Change from Baseline at 24 weeks (V2)，Change from Baseline at 48 weeks (V3)
  use a tweezer to clamp the incisal areas of the anterior teeth or the pit groove on the occlusal surface of the posterior teeth and shake the teeth faciolingually, mesiodistally and vertically I degree : abnormal mobility faciolingually or less than 1mm positioning II degree : abnormal mobility faciolingually and mesiodistally or loosening range of 1-2mm.
  III degree : abnormal mobility faciolingually, mesiodistally and vertically or loosening range is greater than 2mm.
BOP(bleeding of probe) | Baseline(V0)，Change from Baseline at 12 weeks (V1)，Change from Baseline at 24 weeks (V2)，Change from Baseline at 48 weeks (V3)
  observe for 10-15 seconds after probe to see whether it bleeds.Record six sites of each tooth (the mesial, median and distal site of the buccal and tongue surface ).
RBL（adiographic bone level） | Baseline(V0)，Change from Baseline at 24 weeks (V2)，Change from Baseline at 48 weeks (V3)
  Locate the reference point at the deepest PD site of the affected tooth：cemento-enamel junction（CEJ），alveolar crest（AC），bone defect（BD）.RBL is the straight line distance from CEJ to BD (mm)
IC | Baseline(V0)，Change from Baseline at 24 weeks (V2)，Change from Baseline at 48 weeks (V3)
  IC is the straight line distance from AC to BD (mm)
regenerated bone volume parameters | Baseline(V0)，Change from Baseline at 24 weeks (V2)，Change from Baseline at 48 weeks (V3)
  in mimics software, threshold was set according to the gray value of the affected tooth and its surrounding alveolar bone, image editing and region growth were used to form a mask of the three-dimensional reconstruction area. The three-dimensional calculation function was used to reconstruct the three-dimensional shape of the alveolar bone in the target area. Furthermore, the structure of alveolar bone was optimized by remeshing and smooth. The volume of alveolar bone before and after operation was calculated by Boolean operation to obtain the model of regenerated alveolar bone and its volume was measured.
Defect fill (%) | Baseline(V0)，Change from Baseline at 24 weeks (V2)，Change from Baseline at 48 weeks (V3)
  Defect fill (%) = (preoperative IC- and postoperative IC) / preoperative IC × 100%
Defect resolution (%) | Baseline(V0)，Change from Baseline at 24 weeks (V2)，Change from Baseline at 48 weeks (V3)
  Defect resolution (%) = (preoperative RBL- and postoperative RBL) / preoperative RBL × 100%

CONTACTS AND LOCATIONS:
Locations (1):
- Lei Lihong, Hangzhou, China

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-11-19): https://cdn.clinicaltrials.gov/large-docs/60/NCT04953260/Prot_SAP_000.pdf
  • Informed Consent Form (2020-11-19): https://cdn.clinicaltrials.gov/large-docs/60/NCT04953260/ICF_001.pdf